CLINICAL TRIAL: NCT01992471
Title: Multiplex Testing for Breast Cancer Susceptibility: A Pilot Study of Subject Preferences for Information and Responses After Testing
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-215
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: BRCA1 testing; BRCA2 testing; 13-215
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample

GROUPS / COHORTS (1):
- history of breast cancer who have undergone BRCA1/2 testing: This is a single-arm observational study. Subjects with a history of breast cancer who have undergone BRCA1/2 testing and have received uninformative findings will enroll in this study, and then receive pre-test counseling for multiplex testing.
  Interventions: Behavioral: Pre-test Assessment; Behavioral: Pre test Counseling; Other: Blood draw; Behavioral: Post-test counseling, and post-test assessment; Behavioral: Follow-up assessments (6 and 12 months)

INTERVENTIONS:
Behavioral: Pre-test Assessment — Subjects who consent to the study will complete a pre-test instrument that elucidates their baseline response to genetic testing (BRCA1/2) as measured by the Multidimensional Impact of Cancer Risk Assessment (MICRA), and their current cancer surveillance and prevention behaviors, as well asintentions to undergo surveillance and prevention in the next 6 months. The instrument will either be completed at the time of the counseling for multiplex testing, or by phone within approximately 7 days of sample donation.
Behavioral: Pre test Counseling — Subjects will receive appropriate pre-test counseling that will describe the range of outcomes that may results from the multiplex testing. The subject will be asked for permission to audiotape the session for later qualitative review. An outline of the pretest counseling that will be provided. In addition to a description of the genes and syndromes being tested, subjects will receive specific education regarding the following categories and subcategories of possible results a. Definitive (informative) results, b. Variants of uncertain clinical significance (VUCS), c. Uninformative negative test results, d. d. Incidental results. Then Post-counseling selection of desired information After counseling, subjects will complete an instrument indicating which genetic test results they wish to receive. They will complete this instrument in the presence of a genetic counselor, so that the subject may ask questions in order to make the choice most consistent with their preferences.
Other: Blood draw — After choosing the information they wish to receive, subjects will provide a blood sample (2 x 7 cc EDTA tubes, which will be sent to Myriad Genetics Laboratory for analysis.
Behavioral: Post-test counseling, and post-test assessment — When results are available, subjects will be asked to return for in-person communication of the results. Results will be disclosed after confirmation of information preferences in a standard genetic counseling session.
Behavioral: Follow-up assessments (6 and 12 months) — At 6 and 12 months post-results transmission (+/- 4 weeks), subjects will be contacted by telephone by the study RSA to complete follow-up instruments (Assessments 3 and 4; They will complete, by phone, the MICRA. They will also describe the surveillance and prevention behaviors of the preceding 6 months, and their intentions for the next 6 months. Subjects who express a high degree of distress will be offered referral to the Counseling Service, facilitated by Dr. Hay.

SUMMARY:
The purpose of this study is to find out what kinds of information people would like to receive from a new kind of genetic testing, and how they respond to this new kind of testing.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18 or older
* Personal history of breast cancer AND one of the following:
* Invasive breast cancer or DCIS diagnosed at or before age 45 Invasive breast cancer diagnosed at/before age 50 with one or more of the following:
* Limited family history (Fewer than 2 first- or second-degree female relatives in the same lineage that lived to age 45. The "limited family history" can occur on either the maternal or paternal side of the family.)
* 1 or more first-/second-degree relatives with invasive BC at/before 50
* 1 or more first-/second-degree relatives with invasive epithelial ovarian cancer (any age)
* 1 or more first- or second-degree relatives with male breast cancer
* 2 or more first- or second-degree relatives with pancreas cancer
* Invasive breast cancer diagnosed at or before age 60 with at least 2 first or second-degree relatives affected with any combination of invasive breast cancer before age 50, invasive epithelial ovarian cancer at any age, male breast cancer, or pancreas cancer.
* Full sequence BRCA1 and BRCA2 testing completed with no deleterious mutation identified.

Exclusion Criteria:

* Unable to provide informed consent for testing
* Unable to complete English language questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will also be eligible if they are referred to the MSKCC Clinical Genetics Service from outside providers after receiving negative full sequence BRCA1/2 results from those outside providers.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2013-11; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
women's preferences with respect to the type of information they would like to receive from multiplex testing | 2 years
  Proportions of subjects declaring a pre-test preference to receive 1) all available information, 2) all information related to breast cancer predisposition (whether or not clinical utility is established), 3) all information of established clinical utility (whether related to breast cancer risk or not), 4) only a subset of high-penetrance information (masking certain results), 5) no information.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/